CLINICAL TRIAL: NCT02159729
Title: Long-term Follow-up Study of Subjects Who Completed Kythera-sponsored Trials of ATX-101 (Sodium Deoxycholate Injection) for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Long Term Follow-up Study on Safety and Maintenance of Efficacy of ATX-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ATX-101-08-12
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Submental Fat; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants treated with placebo in previous ATX-101 studies
  Interventions: Drug: Placebo
- ATX-101 (1 mg/cm^2) (Experimental): Participants treated with ATX-101 (1 mg/cm^2) in previous phase 2 studies
  Interventions: Drug: ATX-101 (1 mg/cm^2)
- ATX-101 (2 mg/cm^2) (Experimental): Participants treated with ATX-101 (2 mg/cm^2) in previous phase 2 studies
  Interventions: Drug: ATX-101 (2 mg/cm^2)
- ATX-101 (4 mg/cm^2) (Experimental): Participants treated with ATX-101 (4 mg/cm^2) in previous phase 2 studies
  Interventions: Drug: ATX-101 (4 mg/cm^2)

INTERVENTIONS:
Drug: Placebo — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements and recording adverse events
  Arms: Placebo
Drug: ATX-101 (1 mg/cm^2) — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements and recording adverse events
  Arms: ATX-101 (1 mg/cm^2)
Drug: ATX-101 (2 mg/cm^2) — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements and recording adverse events
  Arms: ATX-101 (2 mg/cm^2)
Drug: ATX-101 (4 mg/cm^2) — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements and recording adverse events
  Arms: ATX-101 (4 mg/cm^2)

SUMMARY:
This was a long-term follow-up study of participants who completed Kythera-sponsored trials of ATX-101 (06-03, 07-07, 09-15)

DETAILED DESCRIPTION:
No study medication was administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who successfully completed a Kythera-sponsored clinical trial of ATX-101 (06-03, 07-07, 09-15)
* Signed informed consent
* Willingness to comply with schedule and procedures of the study

Exclusion Criteria:

* Subjects who have had or are undergoing treatment that may affect the evaluation of the submental area will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, MD, PhD, Study Director — Sponsor GmbH
Locations (20):
- United States (10):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Clinical Testing Center Beverly Hills, Beverly Hills, California
  - Mokusiga, Inc, Beverly Hills, California
  - Plastic & Reconstructive Surgery, San Francisco, California
  - Dermatology Institute of DuPage Medical Group in Naperville, Naperville, Illinois
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Body Aesthetic Research Center, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Research Across America, Plano, Texas
- Australia (4):
  - Mei-Heng Tan, Sydney, New South Wales
  - Skin Centre, AHC House, Benowa, Queensland
  - Southeast Dermatology Belmont Specialist Centre, Carina Heights, Queensland
  - T/AS Dermatology Institute of Victoria, South Yarra, Victoria
- Canada (4):
  - Niagara Falls Dermatology & Skin Care, Niagara Falls, Ontario
  - Institute of Cosmetic & Laser Surgery, Oakville, Ontario
  - Toronto Cosmetic Skin Surgery Centre, Toronto, Ontario
  - Cosmetic Dermatology on Bloor, Toronto, Ontario
- United Kingdom (2):
  - The Dermatology Centre, Salford, Manchester
  - Cranley Clinic, Harcout House, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this non-treatment, placebo-controlled, 5-year follow-up study was to evaluate the long-term efficacy and safety of subcutaneous (SC) injections of deoxycholic acid (ATX-101) in the submental area. No treatment was administered in this study.
Pre-assignment Details: Participants who previously received deoxycholic acid or placebo injections in studies ATX-101-06-03, ATX-101-07-07, & ATX-101-09-15 were enrolled in this non-treatment follow-up study to further evaluate safety and efficacy.
Groups:
- ATX-101 (Deoxycholic Acid) Injection: This is a non-treatment follow-up study. Participants were previously treated with deoxycholic acid injection, 10 mg/mL in 1 of 3 predecessor studies ATX-101-06-03, ATX-101-07-07, and ATX-101-09-15
- Placebo: This is a non-treatment follow-up study. Participants were previously treated with placebo in 1 of 3 predecessor studies ATX-101-06-03, ATX-101-07-07, and ATX-101-09-15
Period: Overall Study
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Started | 140 | 65
Completed | 98 | 44
Not Completed | 42 | 21
Not completed — Adverse Event | 0 | 1
Not completed — Subject's Request | 13 | 10
Not completed — Lost to Follow-up | 24 | 9
Not completed — Non compliance | 2 | 0
Not completed — Other Unspecified | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo | Total
Number analyzed (Participants) | 140 | 65 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Visit 0 (Day 0); date of last visit in the predecessor study to which a participant was originally enrolled.
  Years | 46.8 (8.86) | 48.2 (9.94) | 47.2 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 43 | 154
  Male | 29 | 22 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 131 | 56 | 187
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Baseline weight (kg) [Mean (Standard Deviation); unit: kilogram (kg)] | 80.64 (16.683) | 85.93 (15.983) | 82.32 (16.610)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining CR-SMFRS 1-Grade Response During 5 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: Up to 60 months from long-term follow-up (LTFU) baseline (the last visit in the previous study)
Population: Analysis population included all who received study treatment from a previous study, and who were CR-SMFRS 1-Grade Responders at LTFU Baseline
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 104 | 20
percentage of participants
  Baseline | 100.0 | 100.0
  Visit 1 (Month 3): number analyzed (Participants) | 29 | 6
  Visit 1 (Month 3) | 93.1 | 83.3
  Visit 2 (Month 6): number analyzed (Participants) | 67 | 16
  Visit 2 (Month 6) | 94.0 | 68.8
  Visit 3 (Month 9): number analyzed (Participants) | 79 | 16
  Visit 3 (Month 9) | 94.9 | 81.3
  Visit 4 (Month 12): number analyzed (Participants) | 84 | 17
  Visit 4 (Month 12) | 94.0 | 82.4
  Visit 5 (Month 18): number analyzed (Participants) | 82 | 18
  Visit 5 (Month 18) | 95.1 | 83.3
  Visit 6 (Month 24): number analyzed (Participants) | 77 | 16
  Visit 6 (Month 24) | 89.6 | 75.0
  Visit 7 (Month 36): number analyzed (Participants) | 78 | 17
  Visit 7 (Month 36) | 80.8 | 76.5
  Visit 8 (Month 48): number analyzed (Participants) | 61 | 14
  Visit 8 (Month 48) | 85.2 | 64.3
  Visit 9 (Month 60): number analyzed (Participants) | 73 | 14
  Visit 9 (Month 60) | 71.2 | 71.4

2. Primary Outcome: Percentage of Participants Maintaining PR-SMFRS 1-Grade Response During 5 Years of Follow up, i.e. % of Participants Who Were PR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: Up to 60 months from long-term follow-up (LTFU) baseline (the last visit in the previous study)
Population: Analysis population included all who received study treatment from a previous study, and who were PR-SMFRS 1-Grade Responders at LTFU Baseline
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 41 | 21
percentage of participants
  Baseline | 100.0 | 100.0
  Visit 1 (Month 3): number analyzed (Participants) | 19 | 15
  Visit 1 (Month 3) | 94.7 | 73.3
  Visit 2 (Month 6): number analyzed (Participants) | 34 | 20
  Visit 2 (Month 6) | 94.1 | 80.0
  Visit 3 (Month 9): number analyzed (Participants) | 40 | 18
  Visit 3 (Month 9) | 87.5 | 94.4
  Visit 4 (Month 12): number analyzed (Participants) | 40 | 18
  Visit 4 (Month 12) | 85.0 | 94.4
  Visit 5 (Month 18): number analyzed (Participants) | 36 | 18
  Visit 5 (Month 18) | 80.6 | 83.3
  Visit 6 (Month 24): number analyzed (Participants) | 35 | 17
  Visit 6 (Month 24) | 85.7 | 82.4
  Visit 7 (Month 36): number analyzed (Participants) | 33 | 17
  Visit 7 (Month 36) | 81.8 | 94.1
  Visit 8 (Month 48): number analyzed (Participants) | 32 | 15
  Visit 8 (Month 48) | 78.1 | 80.0
  Visit 9 (Month 60): number analyzed (Participants) | 33 | 15
  Visit 9 (Month 60) | 84.8 | 93.3

3. Primary Outcome: Percentage of Participants Maintaining Composite SMFRS 1-Grade Response During 5 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS and PR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: Up to 60 months from long-term follow-up (LTFU) baseline (the last visit in the previous study)
Population: Analysis population included all who received study treatment from a previous study, and who were composite SMFRS 1-Grade Responders at LTFU Baseline
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 30 | 7
percentage of participants
  Baseline | 100.0 | 100.0
  Visit 1 (Month 3): number analyzed (Participants) | 13 | 4
  Visit 1 (Month 3) | 84.6 | 75.0
  Visit 2 (Month 6): number analyzed (Participants) | 23 | 6
  Visit 2 (Month 6) | 82.6 | 83.3
  Visit 3 (Month 9): number analyzed (Participants) | 29 | 6
  Visit 3 (Month 9) | 82.8 | 100.0
  Visit 4 (Month 12): number analyzed (Participants) | 29 | 7
  Visit 4 (Month 12) | 79.3 | 71.4
  Visit 5 (Month 18): number analyzed (Participants) | 26 | 7
  Visit 5 (Month 18) | 73.1 | 71.4
  Visit 6 (Month 24): number analyzed (Participants) | 26 | 6
  Visit 6 (Month 24) | 73.1 | 83.3
  Visit 7 (Month 36): number analyzed (Participants) | 23 | 7
  Visit 7 (Month 36) | 65.2 | 85.7
  Visit 8 (Month 48): number analyzed (Participants) | 23 | 6
  Visit 8 (Month 48) | 60.9 | 83.3
  Visit 9 (Month 60): number analyzed (Participants) | 23 | 6
  Visit 9 (Month 60) | 73.9 | 83.3

4. Primary Outcome: Percentage of Participants Maintaining Composite SMFRS 2-Grade Response During 5 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS and PR-SMFRS 2-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: as for outcome 3
Time Frame: Up to 60 months from long-term follow-up (LTFU) baseline (the last visit in the previous study)
Population: Analysis population included all who received study treatment from a previous study, and who were composite SMFRS 2-Grade Responders at LTFU Baseline
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 3 | 1
percentage of participants
  Baseline | 100.0 | 100.0
  Visit 1 (Month 3): number analyzed (Participants) | 1 | 1
  Visit 1 (Month 3) | 0.0 | 0.0
  Visit 2 (Month 6) | 66.7 | 100.0
  Visit 3 (Month 9) | 66.7 | 100.0
  Visit 4 (Month 12): number analyzed (Participants) | 2 | 1
  Visit 4 (Month 12) | 100.0 | 100.0
  Visit 5 (Month 18): number analyzed (Participants) | 1 | 1
  Visit 5 (Month 18) | 0.0 | 100.0
  Visit 6 (Month 24): number analyzed (Participants) | 1 | 1
  Visit 6 (Month 24) | 100.0 | 100.0
  Visit 7 (Month 36): number analyzed (Participants) | 1 | 1
  Visit 7 (Month 36) | 100.0 | 0.0
  Visit 8 (Month 48): number analyzed (Participants) | 1 | 1
  Visit 8 (Month 48) | 100.0 | 0.0
  Visit 9 (Month 60): number analyzed (Participants) | 1 | 1
  Visit 9 (Month 60) | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Up to 60 months from the last visit in the previous study
Description: All enrolled participants with a clearly identifiable actual treatment received from a previous ATX-101 study and at least 1 visit in the long-term follow-up (LTFU) study were included in the analysis population. All adverse events (AEs) and serious adverse events (SAEs) that were ongoing at the conclusion of the predecessor Studies ATX-101-06-03, ATX-101-07-07, and ATX-101-09-15, were followed until they resolved or were considered medically stable.
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 1/65
Serious Adverse Events (participants affected / at risk) | 3/140 | 3/65
Other Adverse Events (participants affected / at risk) | 0/140 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection (N=140) | Placebo (N=65)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asymptomatic cystic thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Third degree heart block (Cardiac disorders) | 1 (1) | 0 (0)
Patient died of pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thyroid cancer (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.